CLINICAL TRIAL: NCT06725368
Title: Carboplatin + Paclitaxel + Cetuximab (PCC) After Failure of Pembrolizumab +/- First-line Chemotherapy in Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck: CARPACCIO (CARboplatin PAClitaxel Cetuximab IO Immuno-oncology)
Brief Title: Carboplatin + Paclitaxel + Cetuximab (PCC) After Failure of Pembrolizumab +/- First-line Chemotherapy in Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Acronym: CARPACCIO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-006
Record Dates: First submitted 2024-11-28; First posted 2024-12-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm, prospective, multicenter, open-label phase II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCC (Experimental)
  Interventions: Drug: PCC

INTERVENTIONS:
Drug: PCC — PCC protocol (Paclitaxel - Carboplatin - Cetuximab) by intravenous injection for 16 cycles. 1 cycle lasts 1 week. The Carboplatin + Paclitaxel administration schedule 3 weeks out of 4, with weekly Cetuximab is authorized.
  After 16 cycles: maintenance with Cetuximab 500 mg/m2 every 14 days until unacceptable toxicity or progression or death.

SUMMARY:
This study targets an adult population of patients with recurrent or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC), who have failed after a first line of treatment with pembrolizumab associated or not with chemotherapy and having an indication for a second line of treatment. Patients will be recruited in France in medical oncology departments.

The main objective is to evaluate the objective response rate of PCC in patients with HNSCC with locoregional and/or distant 2nd line metastatic disease after failure of pembrolizumab +/- chemotherapy. The secondary objectives of the study are to evaluate other efficacy parameters by monitoring the progression of the disease, the tolerance of the treatment by collecting adverse effects and quality of life.

The duration of participation in the research is 12 months.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is the 7th most common cancer worldwide.

First-line treatment was shaken up in 2019 by showing that a combination of platinum, 5-fluorouracil (5-FU) and the anti-cell death program-1 (PD-1) immunotherapy, pembrolizumab, improved significantly improved overall survival (OS) compared to the standard EXTREME regimen (platinum, 5-FU and cetuximab).

After this first line and in the absence of a randomized therapeutic trial, the therapeutic strategy is not known. Possible chemotherapies are paclitaxel or methotrexate.

Systemic treatment is indicated for patients with locoregional recurrence not eligible for radiotherapy or surgery with curative intent, or progression of distant metastatic disease.

Cetuximab is approved as a second-line treatment in the United States. For patients whose tumor progresses on pembrolizumab maintenance therapy with a platinum-free interval of at least 3 months, restarting platinum therapy is potentially effective. The combination of platinum with cetuximab and paclitaxel is then possible and potentially more effective than monotherapy, including in fragile patients.

The use of cetuximab in the second line appears all the more interesting since its use immediately after anti-PD-1 immunotherapy gives hope for a form of potentiation, as has been reported in several publications since 2020.

Very recently, the results of a French retrospective study evaluating the effectiveness of chemotherapy based on taxane + cetuximab +/- platinum in 99 patients with HNSCC tumor progression and locoregional or metastatic recurrence after immune checkpoint inhibitors was presented by the team of Peers from the Gustave Roussy Institute. They suggest that this combination was effective in this situation and deserved further investigation.

The only existing prospective study was reported during ASCO meeting in 2023. The Japanese team evaluated in a Phase II trial the efficacy of combining paclitaxel with cetuximab in 35 patients with R/M HNSCC after platinum-based chemotherapy and anti-PD1 immunotherapy. The ORR was 69.7%. The median progression-free survival was 5.6 months, and the overall survival was 13.4 months.

A multicenter retrospective study was presented at ESMO 2023. It analyzed the efficacy of paclitaxel alone (69 patients) and the combination of paclitaxel with cetuximab (83 patients) in patients with R/M HNSCC refractory to platinum-based chemotherapy, taxane-naive, and progressive under immune checkpoint inhibitors. An increase of ORR was assessed for the combination of paclitaxel and cetuximab. The median progression-free survival was 4.9 months, and the overall survival was 9.4 months.

Finally, in a study investigating the efficacy of paclitaxel and cetuximab in 57 patients with R/M HNSCC after failure of first-line treatment including an immune checkpoint inhibitor, the ORR was 47.4%. The median duration of response was 5.5 months and disease control was achieved in 42 patients, resulting in a DCR of 71.9%. The median PFS was 5.9 months and the median OS was 14.0 months. The 6-month PFS and OS rates were 48% and 74%, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years at inclusion
2. Cytological or histological confirmation of the diagnosis of invasive squamous cell carcinoma of the head and neck
3. One of the following locations: oral cavity, oropharynx (known p16 status), larynx or hypopharynx
4. Cancers of unknown primary (CUP) of the head and neck are accepted
5. Metastatic (stage IVc) or recurrent disease in patients ineligible for curative surgical treatment or radiotherapy
6. Indication of a 2nd line after pembrolizumab +/- chemotherapy
7. Chemotherapy-free interval ≥ 3 months
8. ECOG Performance Index (Performance Index) of 0, 1 or 2
9. Patient with a life expectancy of at least 12 weeks
10. Documented progression of a measurable tumor target according to RECIST 1.1
11. Correct biology
12. Patient (male or female of childbearing potential) using a highly effective contraceptive method
13. Willingness and ability to comply with the visit schedule, treatment regimens, examinations and other procedures planned in the study
14. Patient enrolled in a health insurance plan or beneficiary of such a plan
15. Signed informed consent obtained before inclusion (after giving clear, fair and appropriate information)

Exclusion Criteria:

1. Other histology
2. Nasal, paranasal and nasopharyngeal cavities
3. Symptomatic or active brain parenchymal metastases or leptomeningeal tumors
4. Grade ≥2 neuropathy
5. Patients may have previously received radiotherapy. A minimum period of 2 weeks is necessary between palliative or analgesic radiotherapy and the start of treatment
6. Clinically significant heart disease or congestive heart failure NYHA (New York Heart Association) class 2 or greater. Patients must not have had unstable angina (symptoms of angina at rest) or new angina in the last 3 months or myocardial infarction in the last 6 months.
7. History of other primary malignancies, except curatively treated malignancies with no evidence of recurrence, within 3 years before the first dose of treatment and a low potential risk of recurrence or non-recurrent skin cancer. melanoma or lentigo maligna properly treated without evidence of disease or carcinoma in situ adequately treated without evidence of disease. A history of T1 grade bladder cancer or T1 grade kidney cancer is accepted. Cervical carcinoma in situ or breast cancer in situ are accepted. Patients with papillary thyroid carcinoma, basal cell skin carcinoma are accepted. A history of prostate cancer is allowed if it is less than or equal to stage T2N0M0 and a Gleason score of 6.
8. Known hypersensitivity to the active substance or excipient of the treatments under study
9. Any uncontrolled intercurrent pathology
10. Any psychiatric illness/social situation that may limit compliance with study procedures or prevent the patient from giving written informed consent
11. Any chemotherapy or radiotherapy performed within 4 weeks of the first dose of study drug, except palliative radiotherapy to a non-target lesion
12. Major surgery within 4 weeks before the first administration of treatment. Local palliative surgery for isolated lesions is tolerated
13. Phenytoin prescribed for prophylaxis
14. Administration of a live attenuated vaccine within 30 days before the first administration of study treatment, as well as during the duration of study treatment and up to 6 months after the last dose of treatment
15. Participation in another clinical trial of an investigational treatment during the 4 weeks preceding the first administration of the study treatment
16. Pregnant or breastfeeding women
17. Women of childbearing potential must have a negative pregnancy test within 72 hours before starting treatment.
18. Patients presenting hemorrhagic tumor
19. History of allergy to red meat or tick bites or positive results of tests for IgE antibodies against cetuximab (α-1-3-galactose)
20. Patient presenting interstitial lung disease
21. History of organ transplant
22. Concomitant treatment with Hypericum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | every 90 days up to 12 months
  Best radiological response according to RECIST 1.1 criteria Number of patients who had an objective response within 12 months CT or MRI (PET scan is not validated for response evaluation) The evaluation is carried out by the investigator.

SECONDARY OUTCOMES:
Progression-free survival | Every 90 days up to 12 months then according to local practices until the date of first documented progression or date of death from any cause or until 5 years, whichever came first
  Progression events (loco-regional progression, metastatic progression or death whatever the cause) will be collected.
Overall survival | From date of treatment initiation until the date of death or lost to follow-up or until 5 years, whichever came first
  The patient's condition (alive, deceased from whatever cause or lost to follow-up) will be collected beyond 12 months of patient participation.
  Patients alive at the time of analysis will be censored on the date of last contact
Response duration | Every 90 days up to 12 months then according to local practices until the date of first documented progression or date of death from any cause or until 5 years, whichever came first
  Time from date of first documented response (complete or partial response) to date of first subsequent progression or death from any cause
Patient Safety | At 12 months
  Incidence of treatment-emergent adverse events, serious adverse events according to CTCAE V5.0 criteria and deaths
Patient Quality of life | every 90 days up to 12 months
  Assessment of all dimensions of EORTC QLQ-C30 questionnaire
Patient Quality of life | every 90 days up to 12 months
  Assessment of difference on specific symptom scales of EORTC QLQ-HN35 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carole PFLUMIO, MD, Principal Investigator — Centre Paul Strauss
Locations (5):
- France (5):
  - Centre hospitalier Régional de Metz-Thionville, Ars-Laquenexy
  - CHU de Besançon, Besançon
  - Centre Hospitalier de Colmar, Colmar
  - Centre Paul Strauss, Strasbourg
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy